CLINICAL TRIAL: NCT01508065
Title: Measuring and Monitoring Blood Glucose Levels Utilizing Non-invasive Blood Glucose Monitoring Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GlucoVista (Industry)
Responsible Party: Sponsor
Other Study IDs: gluco01
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- controlled type one diabetes mellitus.
  Interventions: Device: Glucometer CGM-305

INTERVENTIONS:
Device: Glucometer CGM-305 — The study procedure consists of three days trial. After each experimental day the results of blood glucose level reading from the non-invasive Glucometer CGM-305 will be compared to the reading from several devices, as following: Abbott Freestyle Libre, the hexokinase assay (YSI 2300 STAT Plus) from the venous and the laboratory blood measurements. First day of trial consists of 8-10 hours and is used to calibrate the non-invasive Glucometer CGM-305 for the specific patient. During the second and third days a fasting experiment is performed and consists of 4-6 hours.

SUMMARY:
Adequate glycemic control in patients with Diabetes Mellitus (DM) is a desired therapeutic goal that can be achieved with a true non-invasive device offering the likelihood of continuous glucose monitoring. Currently, glucose is best monitored by measuring capillary blood from the fingertips, from venous/arterial line blood samples and from a daily calibrated Subcutaneous Blood Glucose Monitor (SBGM) which is a source of severe inconvenience and hence, a lack of compliance.

Thus, the need for non-invasive and easy to operate glucose monitoring in DM patients for strict glycemic control cannot be overemphasized.

The Glucometer CGM-305 blood glucose readings are accurate and measure blood glucose with an acceptable mean relative error when compared to acceptable invasive blood glucose measurements.

The primary objectives of the trial are to determine:

1. The safety of the Glucometer CGM-305 in evaluating blood glucose levels
2. The accuracy of the Glucometer CGM-305 in evaluating blood glucose levels

ELIGIBILITY:
Inclusion criteria:

* Type 1 Diabetic patient.
* Ages: 18 to 65.
* Signed informed consent.
* HbA1c of 6%-9% at screening.
* Males- not involved in active military duty.
* Females-non-child bearing potential or females of child-bearing potential who have a negative pregnancy test (HCG in blood or urine) within 72 hours of informed consent.

Exclusion criteria:

* Active systemic or local infection.
* Any medical condition that, by the investigator judgment, will increase the risk from Hyper and Hypo-Glycemic experiment: seizures, heart disease, hypoglycemia unawareness etc.
* History of malignancy, radiotherapy, or chemotherapy for malignancy (except BCC of the skin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will include subjects with controlled type one diabetes mellitus.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Glucometer CGM-305 blood glucose readings as evaluated by mean relative error when compared to venous blood glucose measured by a laboratory device. | will be assessed after second experimental day
Accuracy of the Glucometer CGM-305 blood glucose readings as evaluated by correlation with values measured by glucose hexokinase based assay | will be assessed after second experimental day
Accuracy of the Glucometer CGM-305 blood glucose readings as evaluated by Clark error grid with measurements of venous blood as the comparing value | will be assessed after second experimental day

SECONDARY OUTCOMES:
The safety of the Glucometer CGM-305 in evaluating blood glucose levels | The study consists of three days trial, first day lasts an 8-10 hours, second and third days last 4-6 hours.
  Safety will be evaluated in a descriptive manner by recording all adverse events in the patient population by number and severity.
  The study will evaluate safety by assessing:
  1. Device related adverse events: local and systemic effects of the Glucometer CGM-305 including: redness, burns, pain , or other complications.
  2. General adverse events: Adverse events not directly related to the Glucometer CGM-305 device but are related to the study procedure (i.e clamping), such as: local infection, blood clot, bleeding, hypoglycemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel